CLINICAL TRIAL: NCT05620277
Title: Quantitative Evaluation of the Effect of Dehydration and Rehydration Levels on Tooth Color Using Various Measurement Techniques
Brief Title: Quantitative Evaluation of the Effect of Dehydration and Rehydration Levels on Tooth Color
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200253bK
Record Dates: First submitted 2022-11-02; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Tooth Discoloration
Keywords: Dehydration; Rehydration; Tooth Color; Dental Photography; Color Measurement
MeSH Terms: conditions — Tooth Discoloration; Dehydration

STUDY DESIGN:
Intervention Model Description: 30 patients will be examined for changes in tooth color after dehydration and rehydration stages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Other): 30 patients will be examined for changes in tooth color.
  Interventions: Diagnostic Test: Mobile Dental Photography; Diagnostic Test: Mobile Dental Photography with cross-polarization filter; Diagnostic Test: Mobile Dental Photography with gray reference card; Diagnostic Test: Mobile Dental Photography with cross-polarization filter and gray reference card; Diagnostic Test: Digital Camera; Diagnostic Test: Digital Camera with cross-polarization filter; Diagnostic Test: Digital Camera with cross-polarization filter and gray reference card; Diagnostic Test: Digital Camera with gray reference card; Diagnostic Test: Rayplicker; Diagnostic Test: Rayplicker with gray reference card; Diagnostic Test: Vita Easyshade; Diagnostic Test: Vita Easyshade with gray reference card

INTERVENTIONS:
Diagnostic Test: Mobile Dental Photography — Tooth color changes of 30 patients will be evaluated using Mobile Dental Photography
Diagnostic Test: Mobile Dental Photography with cross-polarization filter — Tooth color changes of 30 patients will be evaluated using Mobile Dental Photography with a cross-polarization filter
Diagnostic Test: Mobile Dental Photography with gray reference card — Tooth color changes of 30 patients will be evaluated using Mobile Dental Photography with a gray reference card
Diagnostic Test: Mobile Dental Photography with cross-polarization filter and gray reference card — Tooth color changes of 30 patients will be evaluated using Mobile Dental Photography with a cross-polarization filter and gray reference card
Diagnostic Test: Digital Camera — Tooth color changes of 30 patients will be evaluated using a Digital Camera
Diagnostic Test: Digital Camera with cross-polarization filter — Tooth color changes of 30 patients will be evaluated using a Digital Camera with cross-polarization filter
Diagnostic Test: Digital Camera with cross-polarization filter and gray reference card — Tooth color changes of 30 patients will be evaluated using a Digital Camera with a cross-polarization filter and gray reference card
Diagnostic Test: Digital Camera with gray reference card — Tooth color changes of 30 patients will be evaluated using a Digital Camera with a gray reference card
Diagnostic Test: Rayplicker — Tooth color changes of 30 patients will be evaluated using Rayplicker
Diagnostic Test: Rayplicker with gray reference card — Tooth color changes of 30 patients will be evaluated using Rayplicker with gray reference card
Diagnostic Test: Vita Easyshade — Tooth color changes of 30 patients will be evaluated using Vita Easyshade
Diagnostic Test: Vita Easyshade with gray reference card — Tooth color changes of 30 patients will be evaluated using Vita Easyshade with a gray reference card

SUMMARY:
This study aims to evaluate the dehydration and rehydration changes in teeth over time and the quantitative effect of these changes on natural tooth color in the clinic. In addition, it is aimed to evaluate the effectiveness of different color measuring devices used in color detection in the clinic, the use of cross-polarization filters, and white balance calibration in color evaluation. Clinicians will evaluate the results of the time intervals in which dehydration is effective in detectable levels of color change. Considering the quantitative changes in dehydrated and rehydrated teeth, it will be possible to prevent negative results in restorations.

DETAILED DESCRIPTION:
According to the criteria determined in our study, 30 individuals were repeated with their mouths open for 15 seconds, 1 minute, 2 minutes, 3 minutes, and 5 minutes with a camera, MDP device, and the use of these devices with a cross-polarization filter to determine how dehydration will affect the tooth color. For white balance calibration, all the shots will be taken the same way with the gray reference card, and the color measurements of the teeth will be taken with two different spectrophotometers in the determined parameters. After these measurements, patients will be kept with their mouths closed and tooth color measurements will be taken after 30 minutes and 60 minutes of remineralization. The patients will be called again 24 hours after these procedures the final color measurement will be made and the basic color parameters will be recorded. Spectrophotometric images will be analyzed according to the manufacturer's instructions. The spectrophotometer shall be calibrated and used according to the manufacturer's instructions before each measurement set. In restorative dentistry clinical applications, color selection errors, which are irreversible errors caused by the color changes of the teeth due to dehydration, will be determined in detail in a short time due to dehydration in the teeth, as a result of this clinical study, and with the result of rehydration, the color change levels will be determined in detail. return will be determined. In this way, it is aimed to create a clearer template for physicians based on time in terms of color selection in the clinic. It is aimed to avoid the need for renewal and avoid unnecessary sessions, as color harmony can be achieved in restorations made by considering the color changes of the tooth during dehydration and rehydration periods. Different photographic techniques and colorimeters will also help measure color variations. In addition, the sensitivity of the color detection methods used in our study will be evaluated comparatively, ensuring which method gives more accurate and reproducible results in clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* healthy periodontal tissue
* tooth color in A1, A2, or A3

Exclusion Criteria:

* any systemic diseases
* smoking
* restoration or caries in anterior teeth
* vital and devital bleaching application

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-05 (Actual); Primary Completion 2023-06-05 (Estimated); Study Completion 2024-06-05 (Estimated)

PRIMARY OUTCOMES:
Tooth color measurement | 15 seconds
  tooth color changes after 15 seconds (dehydration) will be evaluated using Mobile Dental Photography, Digital Camera, Vita Easyshade and Rayplicker

SECONDARY OUTCOMES:
Tooth color measurement | 1 minute
  tooth color changes after 1 minute (dehydration) will be evaluated using Mobile Dental Photography, Digital Camera, Vita Easyshade and Rayplicker

OTHER OUTCOMES:
Tooth color measurement | 2 minutes
  tooth color changes after 2 minutes (dehydration) will be evaluated using Mobile Dental Photography, Digital Camera, Vita Easyshade and Rayplicker
Tooth color measurement | 3 minutes
  tooth color changes after 3 minutes (dehydration) will be evaluated using Mobile Dental Photography, Digital Camera, Vita Easyshade and Rayplicker
Tooth color measurement | 5 minutes
  tooth color changes after 5 minutes (dehydration) will be evaluated using Mobile Dental Photography, Digital Camera, Vita Easyshade and Rayplicker
Tooth color measurement | 30 minutes
  tooth color changes after 30 minutes (rehydration) will be evaluated using Mobile Dental Photography, Digital Camera, Vita Easyshade and Rayplicker
Tooth color measurement | 60 minutes
  tooth color changes after 60 minutes (rehydration) will be evaluated using Mobile Dental Photography, Digital Camera, Vita Easyshade and Rayplicker
Tooth color measurement | 24 hours
  tooth color changes after 24 hours (rehydration) will be evaluated using Mobile Dental Photography, Digital Camera, Vita Easyshade and Rayplicker

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Haciali, DDS, Principal Investigator — Marmara University Faculty of Dentistry Department of Restorative Dentistry
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after the publication of the article.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: data will be available in 2 years.
Access Criteria: all researchers may access the data of this study